CLINICAL TRIAL: NCT06298253
Title: Behavioral Economics to Implement a Traffic Light Nutrition Ranking System in a Network of Food Pantries: Study 2
Brief Title: Behavioral Economics to Implement a Traffic Light Nutrition Ranking System: Study 2
Acronym: BeWell
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Anne N. Thorndike, MD, MPH, Associate Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024P000832
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Food Insecurity; Implementation Science; Diet, Healthy; Behavioral Economics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Behavioral economics-enhanced SWAP implementation strategy (Experimental): Pantries assigned to the intervention group will receive behavioral nudges for implementing the SWAP nutrition program. These include: 1) invoice labeling with the food labeled as red, yellow, or green; 2) receipt of the SWAP toolkit at no cost; 3) pantry learning communities; 4)incentives to purchase SWAP implementation materials (e.g., shelves); 5) food bank recognition for SWAP implementation.
  Interventions: Behavioral: Behavioral economics-enhanced SWAP implementation
- Basic SWAP implementation strategy (Active Comparator): Pantries assigned to the control arm will receive email communication from the food bank dietitian providing them with information about SWAP, online links to SWAP implementation guides, and encouragement to purchase SWAP Toolkits on their own.
  Interventions: Behavioral: Basic SWAP implementation

INTERVENTIONS:
Behavioral: Behavioral economics-enhanced SWAP implementation — Intervention will include behavioral nudges at baseline and over 12 months to promote use of the SWAP nutrition program for pantries.
  Arms: Behavioral economics-enhanced SWAP implementation strategy
Behavioral: Basic SWAP implementation — Intervention will include basic information about the SWAP program and encouragement to obtain SWAP toolkits.
  Arms: Basic SWAP implementation strategy

SUMMARY:
This is a cluster randomized controlled trial of 30 food pantries affiliated with the Greater Boston Food Bank to test the use of behavioral economics (BE) tools to encourage food pantries to implement the Supporting Wellness at Pantries (SWAP) program, with the goal of fostering accurate use of SWAP traffic light labels on pantry shelves and increasing the healthfulness of foods chosen by pantry clients. Primary outcomes will be assessed at 6 and 12 months to compare the implementation and effectiveness of the SWAP program in the intervention vs. control pantries.

DETAILED DESCRIPTION:
This study will test the use of behavioral economics (BE) tools to encourage food pantries to implement the Supporting Wellness at Pantries (SWAP) program, with the goal of encouraging pantries to use SWAP traffic light labels on pantry shelves and increase the healthfulness of foods chosen by pantry clients. The study design is a 12-month cluster RCT of 30 Greater Boston Food Bank partner pantries comparing a basic SWAP implementation strategy (control, n=15) with a BE-enhanced SWAP implementation strategy (intervention, n=15). Primary outcomes assessed at 6 and 12 months will be implementation of the SWAP program within pantries and improvement of client food choices and dietary quality. At the end of 12 months, the BE-enhanced SWAP implementation strategy will be adapted, updated, and offered to the 15 pantries assigned to control (waitlist) at baseline. The 15 intervention pantries will be followed without further intervention.

ELIGIBILITY:
Inclusion Criteria:

* Food pantries enrolled in the study will be partner agencies of the Greater Boston Food Bank that are maximum client choice, are located within approximately 1 hour driving time of Boston (for logistical feasibility), and are not actively using traffic-light nutrition ranking.
* Food pantry clients that complete assessments must be 18 years or older and speak English or Spanish.

Exclusion Criteria:

* Food pantries that are not affiliated with the Greater Boston Food Bank and are not maximum client choice.
* Food pantry clients that do not speak English or Spanish.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3750 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Pantry SWAP implementation | 6 months and 12 months
  Proportion of pantries in the intervention vs. control group that implement SWAP (e.g., traffic-light labels on shelves)
Percent items (by weight) ordered by pantry that are labeled green or red | 6 months and 12 months
  Using data collected from the food bank ordering platform, this outcome will be the proportions (by weight) of the overall orders from GBFB that are green-labeled and red-labeled according to SWAP ranking categories
Percent of pantry clients' selected food that is green or red | 6 months and 12 months
  Using pantry client basket assessments, the total proportion (by weight) of food selected by the client that is labeled green (or red) will be calculated for each participant
Client dietary quality score | 6 months and 12 months
  Rapid Prime Dietary Quality Score (range 0 to 52, higher is healthier) collected at the time clients are leaving the pantry

SECONDARY OUTCOMES:
Skin carotenoid level | 6 months and 12 months
  Measured using the Veggie Meter scale at the time clients leave the pantry; range is 0 to 800 units, with higher scores indicating higher carotenoid levels (and therefore higher fruit and vegetable intake)

CONTACTS AND LOCATIONS:
Overall Officials: Anne N Thorndike, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Data collected from pantry client assessments at baseline, 6 months, and 12 months will be shared. This includes de-identified survey data, including dietary score data, client basket data with food identified as green, yellow, or red-labeled, and skin carotenoid levels. De-identified and aggregated food pantry ordering data, which is secondary data collected from the food bank ordering, will also be shared. The data and details related to our analytic plan and study measures will be deposited in a publicly accessible data repository, such as the Harvard Dataverse, a NIH-approved Scientific Generalist Data Repository free to researchers inside and outside of the Harvard community.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Analytic plans and details will be made available no later than the official publication date of a peer-reviewed article and will be available for at least five years after the study period ends. De-identified data from the study will be made publicly available through the data repository within 90 days of the closeout of the project and made available according to the Harvard Dataverse's data retention policy. Additionally, data for each publication will be deposited by the time of publication.
Access Criteria: In accordance with the data repository methods, completion of a data use agreement form, that stipulates data sharing under an IRB-approved protocol, will be required for accessing the data.

REFERENCES:
- [Derived] Perez PD, Faulkner KC, Wu Y, Schwartz MB, Caspi C, Burgun R, Ortiz L, Jia J, Cheng J, Chang Y, Levy DE, Thorndike AN. Behavioural economics intervention to implement a nutrition ranking system in food pantries: Be Well cluster randomised controlled trial protocol. BMJ Public Health. 2025 Dec 30;3(2):e003650. doi: 10.1136/bmjph-2025-003650. eCollection 2025. PMID 41496767